CLINICAL TRIAL: NCT00909402
Title: Phase 1b Multiple Ascending Dose Study of BMS-833923 (XL139) Administered in Combination With Cisplatin and Capecitabine as First-Line Therapy in Patients With Inoperable, Metastatic Gastric, Gastroesophageal, or Esophageal Adenocarcinomas
Brief Title: A Study of BMS-833923 With Cisplatin and Capecitabine in Inoperable, Metastatic Gastric, Gastroesophageal, or Esophageal Adenocarcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA194-004; 2010-018743-33 (EudraCT Number)
Record Dates: First submitted 2009-05-22; First posted 2009-05-28 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — BMS-833923; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental)
  Interventions: Drug: BMS-833923; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: BMS-833923 — Capsule, Oral, Starting dose 30 mg, Once daily, continuous until discontinuation from study
Drug: Cisplatin — Vial, intravenous (IV), 80 mg/m² IV, Once every 21 days, 1 day per cycle until discontinuation from study
  Other Names: Platinol-AQ
Drug: Capecitabine — Tablets, Oral, 1000 mg/m², twice a day (BID), 14 days per cycle, until discontinuation from study
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of BMS-833923 administered in combination with Cisplatin and Capecitabine as first-line therapy in subjects with inoperable metastatic gastric, gastroesophageal or esophageal adenocarcinomas.

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Esophageal, gastric, or gastroesophageal adenocarcinoma that has spread and cannot be treated with surgery. The diagnosis must be confirmed by a trained pathologist.
* Prior radiation therapy is allowed in certain circumstances - discuss with your doctor.
* Individuals who have had surgery may be eligible after recovering from the procedure.
* Individuals who have received chemotherapy for the treatment of their disease within the past 6 months are not eligible. Chemotherapy given more than 6 months ago is permitted.
* Individuals with spread of their cancer to the brain are permitted in certain circumstances - talk with your doctor.

Exclusion Criteria:

* Significant heart disease.
* Women pregnant or breastfeeding.
* Women able to bear children who are unwilling or unable to use an acceptable method to avoid pregnancy.
* Uncontrolled medical condition or active infection
* Inability to swallow pills.
* Inability to undergo a blood draw, in which a needle is used to obtain blood from a vein in your arm.
* Individuals receiving another drug not approved by the Food and Drug Administration (FDA) or similar agency in another country.
* Prisoners or individuals currently receiving treatment for a mental or physical illness as an inpatient in a hospital.
* Individuals who have experienced pancreatitis, an inflammation of the pancreas, in the past, or who have had a computed axial tomography (CT) scan showing pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Use National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) to establish the MTD, Dose Limiting Toxicity (DLT(s)) and safety profile of BMS-833923 administered in combination with Cisplatin and Capecitabine | At a minimum on days 1, 8, 15 and 35 of cycle 1, days 1 & 14 for cycle 2 and every 21 days thereafter
  MTD - maximum tolerated dose

SECONDARY OUTCOMES:
To evaluate the safety of single-agent BMS-833923, by assessing the evaluation of number, character and duration of adverse event (AE)/serious adverse event (SAE)s | At a minimum on days 1, 8, 15 and 35 of cycle 1, days 1 & 14 for cycle 2 and every 21 days thereafter
Pharmacodynamic effects of BMS-833923 will be measured in tumor biopsy samples taken prior to and during single-agent and combination treatment by evaluation of protein or mRNA of biomarkers of Hedgehog (HH) pathway activation, such as GLI-1 | During cycle 1
  Glioma-associated oncogene (GLI)
  mRNA - messenger Ribonucleic acid
Pharmacodynamic effects of BMS-833923 will be measured in tumor biopsy samples taken prior to and during single-agent and combination treatment by evaluation of protein or mRNA of biomarkers of Hedgehog (HH) pathway activation, such as GLI-1 | During cycle 2
  Glioma-associated oncogene (GLI)
Pharmacodynamic effects of BMS-833923 will be measured in tumor biopsy samples taken prior to and during single-agent and combination treatment by evaluation of protein or mRNA of biomarkers of Hedgehog (HH) pathway activation, such as GLI-1 | During cycle 3
  Glioma-associated oncogene (GLI)
The pharmacokinetic parameters that will be assessed include: Cmax (Maximum observed plasma concentration) | During cycles 1, 2 & 3
The pharmacokinetic parameters that will be assessed include: Tmax (Time of maximum observed plasma concentration) | During cycles 1, 2 & 3
The pharmacokinetic parameters that will be assessed include: AUC(TAU) (Area under the concentration-time curve in one dosing interval) | During cycles 1, 2 & 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (3):
  - City Of Hope National Medical Center, Duarte, California
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
- Local Institution, Toronto, Ontario, Canada
- Local Institution, Villejuif, France
- Local Institution, Amsterdam, Netherlands

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx